CLINICAL TRIAL: NCT02093676
Title: Development and Assessment of a Treatment Protocol for Poorly Controlled Diabetic (Type 1) Adolescents, Based on "The New Authority" Model
Brief Title: Applying the "New Authority" Model in the Treatment of Poorly Controlled Diabetic Adolescents and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0770-YRK-CTIL
Record Dates: First submitted 2014-02-27; First posted 2014-03-21 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; type 1; adolescents; parents counselling
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- parents counseling (Experimental): parents counseling guided by the experiment protocol
  Interventions: Behavioral: experimental protocol treatment "The New Authority"

INTERVENTIONS:
Behavioral: experimental protocol treatment "The New Authority"
  Other Names: "The New Authority" model

SUMMARY:
It is presumed that families of poorly controlled diabetic adolescents (type 1) would benefit from parents' counselling, guided by "the New Authority" model.

DETAILED DESCRIPTION:
"The New Authority" model has been shown to be helpful in risk behaviors such as children's violence and school refusal. It is assumed the model would prove helpful in the risk behavior of lack of adherence to diabetes treatment regimen. The treatment is give to parents only, without the adolescent's participation. It is predicted to improve self care, parents' monitoring, family conflict and parents' helplessness.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes type 1
* condition duration a year or more

Exclusion Criteria:

* family does not speak Hebrew
* adolescent doesn't live at home
* serious psychiatric condition in the family

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
change in self monitoring of blood glucose | assessment at 4 points: enrty, after 3 months, after 6 months and after 9 months

SECONDARY OUTCOMES:
change in reported adherence | assessment at four points: entry, after 3 months, after 6 months and after 9 months
  self care inventory questionnaire
change in parents' helplessness | assessment at four points: entry, after 3 months, after 6 months and after 9 months
  parents' helplessness questionnaire
change in family conflict | assessment at four points: entry, after 3 months, after 6 months and after 9 months
  diabetes family conflict scale
change in parental monitoring | assessment at four points: entry, after 3 months, after 6 months and after 9 months
  parental monitoring of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Orit Hamiel, M.D., Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel